CLINICAL TRIAL: NCT04903574
Title: An mHealth Intervention for Sedentary Behavior in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Abbi Danielle Lane-Cordova, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00110591
Record Dates: First submitted 2021-05-14; First posted 2021-05-26 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Related; Sedentary Behavior
Keywords: Pregnancy; Smartphone; mHealth
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary behavior smartphone app (Experimental): This arm will be assigned to download and use a smartphone app that prompts you to stand up when your smartphone detects 30 minutes of sitting.
  Interventions: Behavioral: NEAT!2 sedentary behavior app
- Pregnancy smartphone app (Active Comparator): This arm will download and use a commercially available pregnancy smartphone app that does not attempt to change activity behavior.
  Interventions: Other: Pregnancy smartphone app

INTERVENTIONS:
Behavioral: NEAT!2 sedentary behavior app — This is a smartphone app that reminds you to stand up if you've been sitting for at least 30 minutes.
  Arms: Sedentary behavior smartphone app
Other: Pregnancy smartphone app — This is a commercially available general pregnancy smartphone app
  Arms: Pregnancy smartphone app

SUMMARY:
Pregnancy outcomes, such as excessive gestational weight gain and gestational diabetes, are linked to long and short-term maternal and child health. Interventions aimed at improving health behaviors, such as sedentary behavior (SB; i.e., any behavior in a seated or reclining position with low energy expenditure) are attractive because they are low-cost, can be disseminated in a wide variety of populations once pregnancy begins, and do not require drugs or prescriptions. Studies have linked SB to some pregnancy outcomes. To the investigators' knowledge, no studies have tested the efficacy of an intervention to reduce SB in pregnant women.

Over 90% of reproductive aged women own a smartphone with similar rates of ownership among black, white, and Hispanic/Latina women, and most adults carry smartphones while awake. Smartphones can monitor SB without additional equipment. Thus, smartphones offer a streamlined opportunity to intervene on SB. The purpose of the research is to evaluate the effectiveness and perception of an mHealth intervention aimed at changing SB in pregnant women. Investigators will survey providers regarding their SB opinions and counseling practices

DETAILED DESCRIPTION:
Investigators will recruit 28 pregnant women, 14 per arm, to participate in this pilot randomized, controlled study. Particiants will complete an in-person baseline study visit in early pregnancy (< week 16). The visit will occur in the Public Health Research Center, Discovery Building, or at a Prisma Health facility. Measurements at the in-person visit (~ 1 hr) include demographics, surveys regarding current and pre-pregnancy PA and SB, medical and pregnancy history, height, and weight. All participants will be given an activPAL(TM) (Glasgow, UK) at V1 to objectively measure SB for 1 week using gold-standard methodology. At the end of the 1-week run-in period (i.e., the week during which SB is objectively measured prior to randomization), participants will mail back the activPAL(TM) and be randomized to the mHealth SB intervention or control group for 12 weeks. SB will be objectively measured again using the activPAL(TM) from week 11-12 of the study. Surveys (Nausea and Vomiting of Pregnancy, Global Health Scales, inquiry about new diagnoses) will be administered remotely in week 5 and week 11. A recruitment opinion survey will be administered remotely in week 5 to inform future recruitment efforts. Surveys related to the intervention platform and perceived effectiveness will be administered remotely at week 12 to participants in the experimental group. Investigators will ask about new diagnoses or adverse events at week 5 and week 11. Investigators will link to participants' medical charts and abstract in-clinic body weight, the results of the third trimester glucose tolerance test, and any other pregnancy-related diagnoses. Investigators will survey Ob/Gyn clinicians (doctors, residents, and nurses) regarding their perceptions of SB during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* currently <16 weeks pregnant with a single infant
* at least 18 years old
* normal weight, overweight, or obese body mass index prior to pregnancy
* can read English at a 6th grade level
* planning to continue pregnancy to term
* owns smartphone and keeps it within arms reach during the day
* willing to allow medical chart access for specific information during the current pregnancy
* no absolute contraindications to exercise, i.e., a doctor has not told you not to exercise during pregnancy

Exclusion Criteria:

* pre-pregnancy BMI <18.5 kg/m2
* age <18 years
* gestational age >16 weeks
* multiple gestation
* not planning to continue pregnancy to term
* does not own a smartphone or keep smartphone within arms-reach during the day
* pre-pregnancy type I or II diabetes
* absolute contraindication to PA in pregnancy
* not receiving prenatal care or not willing to allow access to medical chart
* inability to read English at a 6th grade level.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Time spent in sedentary behavior | Week 11-12 of the intervention
  Total minutes/day in sedentary behavior
Weight gain | At delivery
  Pregnancy weight gain
Glucose tolerance test results | At clinic 1 ay visit glucose test
  The blood glucose level at the third trimester glucose tolerance test

SECONDARY OUTCOMES:
Pregnant patients' opinions of sedentary behavior | Baseline (before randomization)
  Survey regarding feelings about sedentary behavior during pregnancy
Pregnant patients' opinions of the NEAT!2 app | Week 12
  Survey regarding feelings about the app for those assigned to the experimental group
Providers' opinions and practices regarding sedentary behavior | until study is completed; about 1 year
  MD/DO, RN, NP opinions and counseling practices related to sedentary behavior in pregnant patients

CONTACTS AND LOCATIONS:
Overall Officials: Abbi D Lane-Cordova, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are willing to share deidentified data with other researchers. Researchers can contact us if they are interested.